CLINICAL TRIAL: NCT04201678
Title: Investigation of the Effectiveness of Erector Spinae Plane Block in Patients Undergoing Kyphoplasty
Brief Title: Effectiveness of Erector Spinae Block in Kyphoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Assistant professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19/341
Record Dates: First submitted 2019-12-04; First posted 2019-12-17 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Spinal Fractures; Anesthesia, Regional; Anesthetics, Local; Analgesia
Keywords: Kyphoplasty; Erector Spinae Block; conventional local infiltration anesthesia; Extrapedicular infiltration anesthesia
MeSH Terms: conditions — Spinal Fractures; Agnosia

STUDY DESIGN:
Intervention Model Description: Patients will be divided into three randomized groups according to anesthetic method with conventional local anesthesia infiltration (CLIA) method and extrapedicular infiltration anesthesia (EPIAA) and US guided erector spina group (ESP).
Who Masked: Participant, Care Provider
Masking Description: participants and healthcare providers will not know which patient is in which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CLIA (conventional local anesthesia infiltration) Group (Active Comparator): The first step was to determine the pedicle to be vertebroplasty, and 5 mL of 1% Lidocaine Hydrochloride bilaterally to infiltrate the skin, subcutaneous tissue and a portion of the lumbodorsal muscles from a point of 1 cm to the pedicle projection point.
  In the CLIA group, the needle (50 mm 22 Gauge) was directed towards the laminar periosteum at the pedicular projection point at the 10-15 ° angle with the sagittal plane. A mixture of 3 mL of 2% Lidocaine Hydrochloride and 7 mL of 0.5% bupivacaine will be applied bilaterally.
  Interventions: Procedure: CLIA Group (conventional local anesthesia infiltration)
- EPIAA (Extrapedicular infiltration anesthesia) Group (Active Comparator): The first step was to determine the pedicle to be vertebroplasty, and 5 mL of 1% Lidocaine Hydrochloride bilaterally to infiltrate the skin, subcutaneous tissue and a portion of the lumbodorsal muscles from a point of 1 cm to the pedicle projection point.
  The anesthesia process of the CLIA + EPIA group also includes the third step called EPIA. For this stage, the anesthetic needle (50 mm 22 Gauge) is first drawn into the subcutaneous tissue, then through the lateral superior articular process to the lateral half of the pedicle and the upper border of the transverse process (5-10 degrees with sagittal plane and 5-10 with coronal plane), and after negative aspiration 3 mL 2% Lidocaine Hydrochloride and 7 mL 0.5% bupivacaine mixture will be applied bilaterally
  Interventions: Procedure: EPIAA Group (Extrapedicular infiltration anesthesia)
- ESP (Erector Spina Plane Block) Group (Active Comparator): The first step was to determine the pedicle to be vertebroplasty, and 5 mL of 1% Lidocaine Hydrochloride bilaterally to infiltrate the skin, subcutaneous tissue and a portion of the lumbodorsal muscles from a point of 1 cm to the pedicle projection point.
  In the ESP group, a high-frequency-50 15-6 Megahertz (MHz) linear ultrasound probe will be placed vertically approximately 3 cm laterally at the point of application. Once the erector spinae muscle and transverse process have been identified, the peripheral nerve blockage needle (50 mm 22 Gauge) will be advanced from caudal to cranial between the fascia of the erector spina muscle and the transverse process. After 1 ml normal saline injection, this plane was opened. Bilateral 3 mL of 2% Lidocaine Hydrochloride and 7 mL of 0.5% bupivacaine will be administered.
  Interventions: Procedure: ESP Group (Erector Spina Block)

INTERVENTIONS:
Procedure: CLIA Group (conventional local anesthesia infiltration) — The first step was to determine the pedicle to be vertebroplasty, and 5 mL of 1% Lidocaine Hydrochloride bilaterally to infiltrate the skin, subcutaneous tissue and a portion of the lumbodorsal muscles from a point of 1 cm to the pedicle projection point.
  In the CLIA group, the needle (50 mm 22 Gauge) was directed towards the laminar periosteum at the pedicular projection point at the 10-15 ° angle with the sagittal plane. A mixture of 3 mL of 2% Lidocaine Hydrochloride and 7 mL of 0.5% bupivacaine will be applied bilaterally.
  Arms: CLIA (conventional local anesthesia infiltration) Group
Procedure: EPIAA Group (Extrapedicular infiltration anesthesia) — The first step was to determine the pedicle to be vertebroplasty, and 5 mL of 1% Lidocaine Hydrochloride bilaterally to infiltrate the skin, subcutaneous tissue and a portion of the lumbodorsal muscles from a point of 1 cm to the pedicle projection point.
  The anesthesia process of the CLIA + EPIA group also includes the third step called EPIA. For this stage, the anesthetic needle (50 mm 22 Gauge) is first drawn into the subcutaneous tissue, then through the lateral superior articular process to the lateral half of the pedicle and the upper border of the transverse process (5-10 degrees with sagittal plane and 5-10 with coronal plane), and after negative aspiration 3 mL 2% Lidocaine Hydrochloride and 7 mL 0.5% bupivacaine mixture will be applied bilaterally
  Arms: EPIAA (Extrapedicular infiltration anesthesia) Group
Procedure: ESP Group (Erector Spina Block) — The first step was to determine the pedicle to be vertebroplasty, and 5 mL of 1% Lidocaine Hydrochloride bilaterally to infiltrate the skin, subcutaneous tissue and a portion of the lumbodorsal muscles from a point of 1 cm to the pedicle projection point.
  In the ESP group, a high-frequency-50 15-6 MHz linear ultrasound probe will be placed vertically approximately 3 cm laterally at the point of application. Once the erector spinae muscle and transverse process have been identified, the peripheral nerve blockage needle (50 mm 22 Gauge) will be advanced from caudal to cranial between the fascia of the erector spina muscle and the transverse process. After 1 ml normal saline injection, this plane was opened. Bilateral 3 mL of 2% Lidocaine Hydrochloride and 7 mL of 0.5% bupivacaine will be administered.
  Arms: ESP (Erector Spina Plane Block) Group

SUMMARY:
As of October 2019, when the investigators received the approval of the ethics committee, patients who were decided to undergo kyphoplasty with vertebral compression fracture will be included in the study. The patients will be divided into three groups according to the anesthetic method as conventional local anesthesia infiltration (CLIA) method and extrapedicular infiltration anesthesia (EPIAA) and 30 other patients as US guided erector spina group (ESP) for a total of 60 patients. The degree of pain in the intraoperative period will be assessed using a numerical rating scale. Patients with severe pain (NRS> 4) will receive 50 micrograms of fentanyl as an additional analgesic. Sedation levels of the patients will be evaluated with ramsey sedation scale (1-6). Patients with a sedation score of 1 will receive 2 mg of midazolam. During the procedure, pain scores at 0 minutes, 15, 30 and 45 minutes, sedation scores, additional analgesic and sedation amounts administered, and hemodynamic parameters will be recorded. The statistical difference between the groups will be compared

DETAILED DESCRIPTION:
After the approval of the Ethics Committee in October 2019, kyphoplasty patients with vertebral compression fractures will be included in the study. Before the procedure, necessary information will be given to the patients and all of the patients will have their consent to work. Patients will be randomized into three groups. According to the anesthetic method, 30 patients will be classified as conventional local anesthesia infiltration (CLIA) method and 30 patients will be classified as extrapedicular infiltration anesthesia (EPIAA) and 30 others will be classified as US guided erector spina group (ESP). All patients will receive 2 mg midazolam before sedation. In all groups, the pedicle will be determined as the first step and 5 mL of 1% Lidocaine Hydrochloride will be applied bilaterally to the skin, subcutaneous tissue and a portion of the lumbodorsal muscles at a point of 1 cm to the pedicle projection point. In the CLIA group, the needle was directed towards the laminar periosteum at the pedicular projection point at the 10-15 ° angle with the sagittal plane. A mixture of 6 mL of 1% Lidocaine Hydrochloride and 14 mL of 0.5% bupivacaine will be applied.

The anesthesia process of the CLIA + EPIA group also includes the third step called EPIA. For this stage, the anesthetic needle is first drawn into the subcutaneous tissue, then through the lateral superior articular process to the lateral half of the pedicle and the upper border of the transverse process (5-10 degrees with sagittal plane and 5-10 with coronal plane), and after negative aspiration 3 mL 1% Lidocaine Hydrochloride and 7 mL 0.5% bupivacaine mixture will be applied bilaterally. In the ESP group, a high-frequency 15-6 megahertz linear ultrasound probe will be placed vertically approximately 3 cm laterally at the point of application. Once the erector spinae muscle and transverse process have been identified, the peripheral nerve blockage needle (50 mm 22 G ) will be advanced from caudal to cranial between the fascia of the erector spina muscle and the transverse process. After 1 ml normal saline injection, this plane was opened. 6 mL of 1% Lidocaine Hydrochloride and 14 mL of 0.5% bupivacaine will be administered. The entire dose of Lidocaine Hydrochloride shall not exceed 300 mg or <4.5 mg / kg. The degree of pain in the intraoperative period will be assessed using a numerical rating scale. Each patient will receive a brief preoperative training to know that NRS 0 is not pain, 10 is maximum pain, and that they will be asked to report their pain using this scale. Patients with severe pain (NRS> 4) will receive 50 micrograms of fentanyl as an additional analgesic. Sedation levels of the patients will be evaluated with ramsey sedation scale (1-6). Patients with a sedation score of 1 will receive 2 mg of midazolam. The sedation level will be aimed at Ramsey 2-3. Hemodynamic assessments during the procedure will be recorded. Mean arterial pressures (mean blood pressure), heart rate and oxygen saturation (SpO2) will be recorded.

During the procedure, pain scores at 0 minutes, 15, 30 and 45 minutes, sedation scores, additional analgesic and sedation amounts administered, and hemodynamic parameters will be recorded. The statistical difference between the groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* The American Society of Anesthesiologists (ASA) score I-III
* 40-80 years old

Exclusion Criteria:

* ASA >III,
* receiving chronic pain treatment
* previous lumbar surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
numeric rating scale (NRS) | NRS pain score at 0. minutes during the kyphoplasty.
  numerical rating pain scale (0 = no pain, 10 = maximum pain to be considered)
numeric rating scale (NRS) | NRS pain scores at 15. minutes during the kyphoplasty
  numerical rating pain scale (0 = no pain, 10 = maximum pain to be considered)
numeric rating scale (NRS) | NRS pain score at 30. minutes during the kyphoplasty.
  numerical rating pain scale (0 = no pain, 10 = maximum pain to be considered)
numeric rating scale (NRS) | NRS pain score at 45. minutes during the kyphoplasty.
  numerical rating pain scale (0 = no pain, 10 = maximum pain to be considered)
ramsey sedation scale (RSS) | RSS score at 0. minutes during the kyphoplasty.
  Ramsay Sedation Scale divides a patient's level of sedation into six categories ranging from severe agitation to deep coma. Level 1: Patient awake, anxious, agitated, or restless, level 2 :Patient awake, cooperative, orientated, and tranquil, Level 3: Patient drowsy, with response to commands Level 4: Patient asleep, brisk response to glabella tap or loud auditory stimulus Level 5:Patient asleep, sluggish response to stimulus, Level 6:Patient has no response to firm nail-bed pressure or other noxious stimuli
ramsey sedation scale (RSS) | RSS score at 15. minutes during the kyphoplasty.
  Ramsay Sedation Scale divides a patient's level of sedation into six categories ranging from severe agitation to deep coma. Level 1: Patient awake, anxious, agitated, or restless, level 2 :Patient awake, cooperative, orientated, and tranquil, Level 3: Patient drowsy, with response to commands Level 4: Patient asleep, brisk response to glabella tap or loud auditory stimulus Level 5:Patient asleep, sluggish response to stimulus, Level 6:Patient has no response to firm nail-bed pressure or other noxious stimuli
ramsey sedation scale (RSS) | RSS score at 30. minutes during the kyphoplasty.
  Ramsay Sedation Scale divides a patient's level of sedation into six categories ranging from severe agitation to deep coma. Level 1: Patient awake, anxious, agitated, or restless, level 2 :Patient awake, cooperative, orientated, and tranquil, Level 3: Patient drowsy, with response to commands Level 4: Patient asleep, brisk response to glabella tap or loud auditory stimulus Level 5:Patient asleep, sluggish response to stimulus, Level 6:Patient has no response to firm nail-bed pressure or other noxious stimuli
ramsey sedation scale (RSS) | RSS score at 45. minutes during the kyphoplasty.
  Ramsay Sedation Scale divides a patient's level of sedation into six categories ranging from severe agitation to deep coma. Level 1: Patient awake, anxious, agitated, or restless, level 2 :Patient awake, cooperative, orientated, and tranquil, Level 3: Patient drowsy, with response to commands Level 4: Patient asleep, brisk response to glabella tap or loud auditory stimulus Level 5:Patient asleep, sluggish response to stimulus, Level 6:Patient has no response to firm nail-bed pressure or other noxious stimuli
Mean Arterial Pressure (MAP) | MAP at 0. minutes during the kyphoplasty.
  mean arterial blood pressures measured noninvasively will be recorded
Mean Arterial Pressure (MAP) | MAP at 15. minutes during the kyphoplasty.
  mean arterial blood pressures measured noninvasively will be recorded
Mean Arterial Pressure (MAP) | MAP at 30. minutes during the kyphoplasty.
  mean arterial blood pressures measured noninvasively will be recorded
Mean Arterial Pressure (MAP) | MAP at 45. minutes during the kyphoplasty.
  mean arterial blood pressures measured noninvasively will be recorded
SpO2 (Oxygen saturation) | SpO2 value at 0. minutes during the kyphoplasty.
  oxygen saturation measured by pulseoximeter will be recorded
SpO2 (Oxygen saturation) | SpO2 value at 15. minutes during the kyphoplasty.
  oxygen saturation measured by pulseoximeter will be recorded
SpO2 (Oxygen saturation) | SpO2 value at 30. minutes during the kyphoplasty.
  oxygen saturation measured by pulseoximeter will be recorded
SpO2 (Oxygen saturation) | SpO2 value at 45. minutes during the kyphoplasty.
  oxygen saturation measured by pulseoximeter will be recorded
Heart rate (HR) | HR at 0. minutes during the kyphoplasty.
  heart rate measured by electrocardiogram will be recorded
Heart rate (HR) | HR at 15. minutes during the kyphoplasty.
  heart rate measured by electrocardiogram will be recorded
Heart rate (HR) | HR at 30. minutes during the kyphoplasty.
  heart rate measured by electrocardiogram will be recorded
Heart rate (HR) | HR at 45. minutes during the kyphoplasty.
  heart rate measured by electrocardiogram will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B EŞKİN, Study Director — Gulhane Training and Research Hospital; Ayşegül Ceylan, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No